CLINICAL TRIAL: NCT03446274
Title: An Open Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-NW-3509 in Healthy Male Subjects
Brief Title: An Open Label, Single-Dose Study of 14C-NW-3509 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NW3509-007
Record Dates: First submitted 2018-01-29; First posted 2018-02-26 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Evenamide — This is an orally available small molecule that potently blocks voltage-gated sodium channels (VGSCs) in vitro and is indicated for the treatment of patients with schizophrenia, mania, and bipolar disorder.

SUMMARY:
This is a single-center, open-label, non-randomized, single dose of 14C-NW-3509 capsule study in 6 healthy male subjects.

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, single dose study in a single cohort of 6 healthy male subjects, including up to 2 cytochrome P450 (CYP)2D6 poor metabolizer subjects. Each subject will receive a single oral administration of 14C-NW-3509 capsule in the fasted state.The screening period and study admission to completion is estimated to be up to 43 days. The following data will be analyzed urine and feces data for total radioactivity, plasma and whole blood data for total radioactivity and plasma concentration data for NW-3509.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
3. Must be willing and able to communicate and participate in the whole study
4. Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day)
5. Subject is considered healthy on the basis of medical history, physical examination, ECG, vital signs and clinical laboratory assessments
6. Must provide written informed consent
7. Must adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Radiation exposure, excluding background radiation but including significant medical exposures, or other trial related exposures, not exceeding 5 mSv in the 12 months preceding participation in the trial, or radiation exposure exceeding 10 mSv in the 5 years preceding participation in the trial, inclusive of the 3 mSv exposure resulting from participation in this study. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study. Significance of a medical exposure will be determined by the investigator.
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
10. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
11. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
13. History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or neurological or psychiatric disorder, as judged by the investigator
14. Presence or history of seizure disorders or ataxia
15. History of presence of significant cardiac conduction abnormalities including but not limited to: PR interval >240 msec; QRS duration >120 msec; QTcF interval >450 msec
16. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
17. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
18. Donation or loss of greater than 400 mL of blood within the previous 3 months
19. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration (See Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
20. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Metabolic profiling for NW-3509 will be determined in plasma, urine and fecal samples | 15 days
  Percent of each radio labeled drug-related material will be determined in plasma, urine and feces

SECONDARY OUTCOMES:
Routes and rate of elimination of NW-3509 in plasma, urine and feces | 15 days
  The routes and rate of elimination of 14C-NW-3509 by measurement of 14C-NW-3509 and its major metabolites in plasma, urine and feces
The identification of major metabolites of NW-3509 in plasma, urine and feces | 15 days
  Metabolic profiling will be performed using liquid chromatography-radio-detection, with subsequent mass spectrometry
Safety and Tolerability of NW-3509 | 15 days
  This will be assessed by Adverse events, Clinical chemistry, Clinical Hematology and Urinalysis, Vital signs and Physical Examination
Oral Pharmacokinetics of NW-3509 in plasma, urine and feces | 15 days
  Several parameters will be measured Cmax, Tmax, AUC, elimination half-life, Tlag etc

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MRCS, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, NG, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided